CLINICAL TRIAL: NCT04065542
Title: Determinants of Health and Cancer: Investigating the Conceptions of Children From 6 to 11 Years Old
Acronym: FCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other)
Responsible Party: Sponsor
Other Study IDs: 2019 FCE
Record Dates: First submitted 2019-05-28; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-05

CONDITIONS: Child; Determinants of Health; Qualitative Research; Cancer
Keywords: Social behaviour; Qualitative research; Child; Cancer
MeSH Terms: conditions — Neoplasms; Social Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Model and map, from a qualitative multi-phased protocol, the conceptions and systems of conceptions of the determinants of health and cancer expressed and perceived by schoolchildren aged 6 to 11 years. The secondary objectives are to analyze the ability to question the conceptions of children's health regardless of their age and to link conceptions and determinants to contextual factors. The informative value and complementarity of the collection tools (photo expression, QC, photo-narration) and the relevance of a mixed analysis methodology (qualitative and quantitative) in order to highlight the different determinants of health will also be studied.

DETAILED DESCRIPTION:
Qualitative observational study of human and social sciences (SHS), multicenter, conducted with schoolchildren.

The qualitative methodology used combines the use of photographs, open questionnaires and focus groups, over very large panels, aiming at both diversity and representativeness.

* Photo expression: to identify the determinants perceived as having a positive or negative influence on one's health;
* CQR : Certainty/Question/Rumour on how to take care of one's health (health promotion input following on from school policies, i.e. PES: Politique d'Etablissements Scolaires);
* Photo narration: to identify argumentative frameworks in health and alternatives perceived as being positive or negative for one's health,
* Focus groups: to improve understanding of the rationalities built by adolescents in relation to that which determines their health.

This choice is justified by the need to explore and understand the actions from the participants' point of view.

The diversity of schools and pupils (5 classes in 4 schools in the AURA region, i.e. 320 pupils) will make it possible to obtain the data saturation required in qualitative research.

This makes it possible to consider a mixed analysis strategy, both qualitative and quantitative.

This project aims to better understand the rationalities elaborated by children and the way in which their concepts on the determinants of cancer interlink, as well as to describe the declared impact these concepts have on the decision-making regarding their health.

ELIGIBILITY:
Inclusion Criteria:

* School volunteering to participate in the project Primary school
* children aged 6 to 11
* Girls and boys
* All school levels Private and public primary school
* Rural and urban primary school

Exclusion Criteria:

* Class ULIS
* Students who benefit from a personalized support plan
* Individual refusal of participation (child and / or family)

Ages: 6 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: chidren
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
categorized groups by genre according to the Relation to the environment criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.
categorized groups by genre according to a Factors of fulfillment and personal development criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.
categorized groups by genre according to the link with a healt theme criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.
categorized groups by genre according to Care activities criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.
categorized groups by genre according to a Recommendation and support in health in the social sphere criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.
categorized groups by genre according to an health capital criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.
categorized groups by genre according to the emotional dimension in social relations criteria | day 1
  The analysis of the content will be carried out according to the ascending / descending method by categorization, described by Laurence Bardin. According to L. Bardin (2013), categorization is an operation of classification of elements constituting a set by differentiation then grouping by genre (analogy) according to previously defined criteria.

SECONDARY OUTCOMES:
Incidence of children able to explain their health regardless of their age | Day 1
  The informative value and complementarity of the collection tools (photo The informative value are measured with collection tools (photo expression, photo-narration) and a mixed analysis methodology (qualitative and quantitative) is used in order to highlight the different determinants of health.
Incidence of children able to explain their health regardless of their contextual factors | Day 1
  The informative value are measured with collection tools (photo expression, photo-narration) and a mixed analysis methodology (qualitative and quantitative) is used in order to highlight the different determinants of health.
Identify child profile | Day 1
  Identify child profiles / classes / school based :• Socio-demographic data (class / age, sex, class size, number of male and female, school enrollment, class number, geographical location, priority education, team stability, health project, type of project, impression of researchers)
  • Domains or designs: Individual & collective Domains created during the qualitative analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Lise LACLAUTRE, Clermont-Ferrand, France